CLINICAL TRIAL: NCT01692067
Title: Combat, Sexual Assault and Post-Traumatic Stress in OIF/OEF Military Women
Brief Title: Deployment Health in Regular Military Women
Acronym: DHRMS
Status: Completed | Type: Observational
Sponsor: Iowa City Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Anne G SAdler, CADRE Core Investigator, Iowa City Veterans Affairs Medical Center
Other Study IDs: PT075819; GRANT00341283 (USAMRMC); DHI08-136 (DVA)
Record Dates: First submitted 2011-07-28; First posted 2012-09-25 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Military Physical and Sexual Trauma; Combat Trauma; PTSD; TBI
Keywords: Rape; Women; Military; Veterans; Post-traumatic Stress Disorder; Traumatic Brain Injury
MeSH Terms: conditions — Sexual Trauma; Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- D0: Not deployed
- D1: Deployed to combat-related regions once
- D2: Deployed to combat related regions more than once
- D3: Deployed outside of the continental US but not to combat related regions

SUMMARY:
The purpose of this study is to determine potential risk factors for physical and sexual assault in regular military women (as opposed to Reserve and National Guard). In addition, this study seeks to determine associations between service women's violence exposures and: current physical and mental health status (e.g. PTSD), and access to and use of DoD, DVA and civilian healthcare.

DETAILED DESCRIPTION:
Background: The proposed study of Regular Military service women builds on and extends a funded VA HSR&D grant currently investigating similar objectives in Reserves and National Guard (R/NG) service women. This proposed study addresses the radically changing DoD and DVA health care delivery needs of two priority populations: women exposed to combat, and women sexually assaulted during military. There is a limited understanding of the complex relationship between these traumatic exposures and women's health outcomes, such as post-traumatic stress disorder (PTSD) and traumatic brain injury (TBI) and with their subsequent health service use or barriers to care.

Objectives: The objectives are: 1) To identify and describe organizational, situational, and individual risk factors for physical and sexual assault (i.e., victimization) in women who have served or are currently serving in the Regular Military in Operation Enduring Freedom and Operation Iraqi Freedom (OEF/OIF) by deployment status (those who are deployed to combat related regions once, those deployed more than once, those serving in non-combat related areas outside of the continental United States (US), or those serving within the continental US. 2) To determine associations between PTSD, TBI, and physical and sexual assault during OEF/OIF with current physical and mental health status and health risk behaviors by deployment status. 3) To identify current internal and external barriers to DoD, DVA, and civilian health services in relationship to women's deployment and victimization status and the association between PTSD and TBI; 4) To identify and describe differences between Regular Military and R/NG populations for each of these objectives.

Methods: We propose a cross sectional study design with two sequential phases. Phase 1 would include focus groups to refine the current study interview specific to Regular Military populations. Phase 2 would involve the identification and successful interviewing of 669 Regular Military service women, using random sampling with stratification by deployment status, state of service accession, and service branch. Building on our current study, women will be selected from five states: Iowa, Illinois, Kansas, Missouri, and Nebraska. Potential study participants will be mailed an information summary and asked to take part in a study assessing the deployment health of military women. 1058 women will be contacted to obtain the target of 669 completed interviews. Consenting participants (167 per deployment group) will complete a telephone interview that assesses socio-demographic variables, trauma exposures, health history, current health status, military environmental factors (organizational and situational factors), military and DVA health care and barriers to this care, and self reported service use. Descriptive analysis and multiple logistic regression analysis will be used.

Implications: It is unclear if the needs of military women are met by current combat-associated PTSD treatments originally based on male populations. It is anticipated that our findings will improve understanding of the health risks and outcomes of deployed Regular Military service women in contrast to women serving in the R/NG (with PTSD and TBI as key outcome variables). Our results consequently will have implications for DoD and DVA evidence based interventions for both primary prevention and care.

ELIGIBILITY:
Inclusion Criteria:

* Focus Group:

  * Men or women who have or are currently active duty regular military (RM) of OIF/OEF service eras (10/7/01- present)
* Interview phase:

  * Women, who have or are currently serving active duty RM during OIF/OEF service eras

Exclusion Criteria:

* Focus Group:

  * Disabilities that render incapable of hearing
  * Comprehending
  * Communicating in a group or inhibit travel to focus group
* Interview phase:

  * Disabilities that render incapable of hearing
  * Comprehending
  * Communicating independently with interviewers by telephone
  * Not having telephone and unable to access a nearby VA or other possible resource to contact toll free number.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women and Men who have or are currently serving in the USA regular military.
Sampling Method: Non-Probability Sample
Enrollment: 871 (Actual)
Dates: Start 2009-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Organizational, situational, and individual risk factors for physical and sexual assault in women who have or currently serving in active duty Regular Military in OIF/OEF by deployment status. | Months 28-42 of grant

SECONDARY OUTCOMES:
Traumatic brain injury | Months 28-42 of grant
Current internal (e.g. PTSD) and external barriers (e.g. access to care factors)to health services | Months 28-42 of grant
Identification and description of differences between Regular Military and Reserve/National Guard service women for each of these aims (building on currently funded grant). | Months 28-42 of grant
PTSD | Months 28-42 of Grant
Current medical health, including reproductive health | Months 28-42 of grant
Deployment factors associated with risk of violence/health | Months 28-42 of grant

CONTACTS AND LOCATIONS:
Overall Officials: Anne G Sadler, Ph.D., Principal Investigator — US Department of Veterans Affairs
Locations (2):
- United States (2):
  - Anne G. Sadler, Ph.D.; VAMC, Iowa City, Iowa
  - Iowa City VAMC, Iowa City, Iowa